CLINICAL TRIAL: NCT06731946
Title: Safety and Efficacy of the Surpass Evolve Flow Diverter in Treating Intracranial Aneurysms
Status: Active, not recruiting | Type: Observational
Sponsor: Yibin Fang (Other)
Responsible Party: Sponsor-Investigator, Yibin Fang, Dr., Shanghai Fourth People's Hospital Tongji University
Organization: Shanghai Fourth People's Hospital Tongji University (Other)
Other Study IDs: SYNXG202401
Record Dates: First submitted 2024-12-11; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Intracranial Arterial Aneurysm
Keywords: Intracranial Arterial Aneurysm; Surpass Evolve Flow Diverter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Surpass Evolve Flow Diverter
  Interventions: Device: Flow diverting

INTERVENTIONS:
Device: Flow diverting — Flow diverter has become the standardized treatment method for Intracranial aneurysms (IAs), which is different from angioplasty, coiling, etc.

SUMMARY:
Safety and Efficacy of the Surpass Evolve Flow Diverter in Treating Intracranial Aneurysms

DETAILED DESCRIPTION:
This study aims to retrospectively evaluate the efficacy and safety of the Surpass Evolve Flow Diverter in treating complex intracranial aneurysms. It seeks to assess long-term outcomes and complication rates while analyzing the impact of patient characteristics and aneurysm types on treatment effectiveness. By collecting data from multiple centers, the study ensures broad representativeness, ultimately providing valuable insights for clinical management on a global scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years with a confirmed diagnosis of intracranial aneurysm.
2. Imaging studies confirming suitability for Surpass Evolve Flow Diverter treatment.
3. Aneurysms meeting flow diverter treatment indications (e.g., aneurysms larger than 4 mm).
4. At least six months of follow-up data available post-treatment.

Exclusion Criteria:

1. Patients with acutely ruptured aneurysms or significant bleeding.
2. Patients with incomplete data or insufficient follow-up records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese populations with intracranial aneurysms
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete aneurysm occlusion rate | 12(-3 ~ +6) months
Favorable prognosis rate | 12(-3 ~ +6) months
  mRS score 0-1
Procedure-related complication rate | 12(-3 ~ +6) months

SECONDARY OUTCOMES:
Procedural success rate | 12(-3 ~ +6) months
Perioperative complication rate | 12(-3 ~ +6) months
Neurological mortality rate | 12(-3 ~ +6) months
Incidence of postoperative stroke/TIA | 12(-3 ~ +6) months
Rates of postoperative intracranial hemorrhage and neurological deficits | 12(-3 ~ +6) months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Fourth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided